CLINICAL TRIAL: NCT04494035
Title: AVATR - Arteriovenous Access Thrombosis Removal With CAPERE Thrombectomy System
Acronym: AVATR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor change
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TP19-0010
Record Dates: First submitted 2020-07-22; First posted 2020-07-31 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Arteriovenous Graft Thrombosis

STUDY DESIGN:
Intervention Model Description: A prospective, single-arm, non-blinded study, intending to treat and collect and evaluate data in up to ten (10) human subjects who are currently being treated with hemodialysis and who present with acute thrombosis in their arteriovenous (AV) grafts, treated with the CAPERE® Thrombectomy System.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- AVATR-Toronto (Experimental): Thrombectomy of arteriovenous graft using CAPERE Thrombectomy System
  Interventions: Device: CAPERE Thrombectomy System

INTERVENTIONS:
Device: CAPERE Thrombectomy System — Arteriovenous graft thrombectomy

SUMMARY:
A prospective, single-arm, non-blinded study, intending to treat and collect and evaluate data in up to ten (10) human subjects who are currently being treated with hemodialysis and who present with acute thrombosis in their arteriovenous (AV) grafts, treated with the CAPERE® Thrombectomy System.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients who are ≥ 18 years of age
* Dialysis patients with clinical signs, symptoms and presentation consistent with acute thrombosis; onset of symptoms ≤ 14 days

Exclusion Criteria:

* Dialysis patients who are ≤ 18 years of age.
* Grafts with aneurysmal degeneration
* Central venous occlusion
* Patients with infection of the vascular access
* Patients with active cancer under current therapy, myeloproliferative syndromes, hyperhomocysteinemia, and heparin-induced thrombocytopenia.
* Patients with pulmonary embolism (PE) with hemodynamic compromise
* Any contraindication to systemic or therapeutic doses of heparin or anticoagulants
* Known anaphylactic reaction of radiographic contrast agents that cannot be pre- treated
* Imaging evidence or other evidence that suggests the participant is not appropriate for mechanical thrombectomy intervention (e.g. recent access site creation where there are concerns of leak or disruption of the suture line)
* Female who is pregnant or nursing
* Concurrent participation in another investigational drug or device treatment study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint (Effectiveness) | Intraoperative
  Clearance of clot and restoration of blood flow within the affected graft as confirmed via angiographic endpoint in conjunction with a clinical or hemodynamic endpoint
Safety Evaluation | 24 Hours
  Aggregated major adverse events of < 5% (events that cannot be adjudicated in less than 24 hours: death, stroke, major bleeding)

SECONDARY OUTCOMES:
Device Safety | Intraoperative
  Successful withdrawal of device along with clots without angiographically significant emboli, vessel trauma, entry site aneurysm, major bleeding complications
Technical Success | Intraoperative
  Ratio of successful thrombus removals and total number of participants
Thrombus Removal Rate | Post-procedure
  Percent of thrombus removal comparing pre-treatment to post-treatment angiography
30-Day Patency Rate | 30-days
  Patency of graft at 30-days post-procedure as assessed by ultrasound or other method
Clinical Success | Open
  Ability to deliver dialysis via the graft post procedure for at least one session

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mafeld, MD, Principal Investigator — University Health Network Toronto General
Locations (1):
- University Health Network Toronto General, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No